CLINICAL TRIAL: NCT03340103
Title: Evaluation of the Antioxidant Activity of Lutein/Zeaxanthin Early Administered to Premature Newborns
Brief Title: Early Administration of the Lutein/Zeaxanthin in Premature Newborns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was not possible
Sponsor: Sooft Italia (Industry)
Collaborators: Fondazione Poliambulanza Istituto Ospedaliero (Other); University of Siena (Other); University Hospital Padova (Other); University Hospital Perugia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3172 10/10/2018
Record Dates: First submitted 2017-10-17; First posted 2017-11-13 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Antioxidant Role of the Lutein in Preterm Newborn
Keywords: Lutein/Zeaxanthin; Antioxidant; Oxidative stress; Carotenoid; Preterm newborn

STUDY DESIGN:
Intervention Model Description: Since birth, premature newborns, that are comply with the inclusion parameters, will be introduced and separated in two random groups (A and B).
  All newborns, during the observation period, will be submitted to the blood collection (1 ml) from the umbilical cord and peripheral site (at the same time with the routine collections) on which there will be performed blood gas analysis and oxidative stress markers (TH and BAP)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pilot study, non-commercial, with food supplement, treated vs. control with a ratio 1: 1 double-blind. The identical vials, corresponding to placebo and active product, have an alphanumeric code without meaning for the operator, but that identifies the treaties from controls, in an anonymous document kept by the Statistical. The document will be placed in a sealed and anonymous envelope and it will be kept open by the statistician at the time of data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): Group A (18 newborns) will be treated with LUTEIN ofta 0,5 drops, (1 ml per Kg equal to 0,5 mg of lutein and 0,05 of zeaxantin) additionaly to the standard hospital treatment foreseen. The first dose will be given within 36 hours of life, the least to 30th day of life.
  Interventions: Dietary Supplement: LUTEIN ofta 0,5 gocce
- Control group B (Placebo Comparator): Group B (18 newborns) treated with Placebo solution additionaly to the standard hospital treatment foreseen. The first dose will be given within 36 hours of life, the least to 30th day of life.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: LUTEIN ofta 0,5 gocce — LUTEIN ofta 0,5 gocce, containing a solution of 5% Lutein and 2,5% Zeaxanthin with excipients (Corn starch, glucose, potassium sorbate, xanthan gum, citric acid)
  Arms: Experimental group A
Drug: Placebo — Placebo solution with unique excipients (Demineralised water, potassium sorbate, xanthan gum, citric acid)
  Arms: Control group B

SUMMARY:
Premature birth is the most common cause of mortality, morbidity and disability. Premature infants have a higher risk of developing damage in the eyes (retinopathy of prematurity ROP), in the central nervous system (intraventricular hemorrhage IVH), in the lungs (bronchial pulmonary dysplasia BPD), in the gut (NEC) and infections. Oxidative stress has been implicated in various capacities, in the etiology of these conditions. Lutein and Zeaxanthin are powerful anti-oxidants and commonly assimilated with different foods. Lutein and Zeaxanthin are present at level of umbilical cord, in the breast milk (particularly in colostrum) and pass the placental barrier. Concerning supplementations, the lutein presents, for its specific characteristics, a high bioavailability after oral administration. In the last few years, there have been more and more studies which have shown that lutein could constitute a valid and important preventive and protective factor against certain diseases related to oxidative stress. The preparations of lutein and zeaxanthin have never pointed out in the human being (included in the term newborn) adverse or toxic effects. This spontaneous / non-commercial pilot study involves the administration of a dietary supplement containing lutein / zeaxanthin, because the healthcare structures need to identify a natural antioxidant product that can reduce the incidence of serious diseases related to oxidative stress in the perinatal period. This study aims to evaluate if the administration of lutein in watery solution will reduce the rate of free radicals in preterm infants.

DETAILED DESCRIPTION:
Lutein is the most important carotenoid present selectively in certain tissues of the human body, mainly at the level of the retina, macula (hence the name) and lens. In tissues and serum, lutein is found together with a carotenoid dihydroxide, its isomer, zeaxanthin. Lutein and zeaxanthin are present at the level of the umbilical cord and pass through the placental barrier and are also present in the plasmatic ones, in breast milk and especially in the colostrum. Concerning the way of administrating, the lutein presents, through its specific characteristics, an elevated bioavailability after oral administration. The hematic levels of lutein, after providing nutriments rich in carotenoids, are increased with 67% from the 14% observed at beta-carotene. Through interdisciplinary and coordinated studies, performed both in vitro and in vivo, there were identified different action mechanisms; particularly, investigators have demonstrated a defense mechanism of the tissue function by lutein, which is produced through the neutralization (quench) phenomenon of the singlet oxygen and reactive oxygen species (ROS). This action provides molecules with different activities: an antioxidant function, anti-inflammatory properties, properties which promote anti-tumoral effects, induction of detoxification enzymes and positive effect on proteins promoting the communication between joints (up-regulation). Recently, there have appeared experimental and chemical data proving that the oxidative stress and harmful actions determined by ROS can play an important role in the pathogenesis of many neurological diseases as Alzheimer, Parkinson in adult and ROP and NEC in newborns.

This is due to the fact that the nervous system is characterized by membranes rich in polyunsaturated fats, the first cellular compounds affected by ROS attack through the lipid peroxidation. A similar mechanism can appear to certain ocular tissues (macula, lens, retina) which, containing high amounts of polyunsaturated fat acids, are more vulnerable than other structures with oxidative degradations induced by ROS.

Due to the fact that carotenoids are amongst the most powerful antioxidants existing in nature, there are being developed new researches concerning the functional role of these substances in preventing neurodegenerative diseases in newborns.

Because these polyunsaturated fat acids are very sensitive to oxidation, the modification of their plasmatic levels influences the state of the antioxidant systems on the mother and subsequently to the foetus. Many studies have proved that the increase of the susceptibility to the peroxidation of polyunsaturated fat acids on pregnant women is accompanied by an equivalent increase of the tocopherol plasmatic concentration which, immediately after birth, decrease sharply.

The plasmatic concentrations of the newborns' antioxidants were lower than those of the mothers. In the umbilical cord, the levels of tocopherols and carotenoids are significantly lower than the ones registered in the maternal plasma and the concentration of polyunsaturated fat acids on the newborn is significantly higher and a lot more increased than on the mother.

Furthermore, specific studies showed a growing interest towards the oxidative stress and oxygen reactive species which supposedly accumulate after birth. Many practices usually used in the delivery room (for example the drugs given to pregnant woman to ease her pain, the newborns' extraction methods, the techniques to minimize body temperature decrease, blocking the umbilical cord and especially the use of oxygen to 100 % or a ventilated room for newborns presenting asphyxia signs) do not always prove to be efficient and can also compromise the health of the newborn because of a significant increase of free radicals.

Some specific studies have compared the levels of free radicals, highlighted with markers, in the plasma of the umbilical cord of newborns with asphyxia treated 100% with oxygen or 21% with oxygen, comparative to a control group of children without asphyxia. The levels of free radicals were significantly increased immediately after birth in all three groups and grew in the two groups of newborns with asphyxia. In the group treated 21% with oxygen, these values decreased and have reached the same level of the newborns without asphyxia at 28 days after birth, whereas at the group treated 100% with oxygen the levels of free radicals remained very high.

Thus, a short exposure of the newborn to 100% oxygen is the cause of an extended oxidative stress state and a consistent increase of free radicals, which seem to be involved in different diseases and pathologies during the first months of life, especially in the preterm infant increasing significantly the incidence of ROP, IVH, BPD, NEC and infections.

These results show that the newborn need to increase the level of antioxidant protection to establish the redox balance and to prevent the problems occurred from an extended exposure to high levels of free radicals and oxygen reactive species.

The premature birth is the most frequent cause of mortality, morbidity and disability. Premature babies have an extremely high risk to develop ocular or neurological lesions. The main complication at visual level that may appear is called retinopathy of prematurity, so called ROP. Oxidative stress is involved in the etiology of this disease. In fact, premature babies, because of respiratory issues, are often exposed to potentially damaging oxygen concentrations or to phototherapy with high blue light intensity. These therapeutic practices are sources of free radicals.

The studies performed on the babies showed that the levels of carotenoids in the first four / six months of life are much reduced. This is due to the fact that the baby's diet is based exclusively on milk, without any solid elements (as vegetables or green leaves), sole sources of this nutrient. Nevertheless, breastfed babies, in average, present high plasmatic lutein levels than babies fed with prepared milk. Different milk formulas for newborns found at present time on the market are not enriched with this type of carotenoids, thus their content of lutein and zeaxanthin is very low, except certain formulas which are not traded in Italy and prepared using egg mixes. Breast milk, is thus the only source of lutein for the newborn before weaning, and breast feeding proves to be of considerable importance as primary source of these micronutrients for the newborn, proper development and visual function protection. Taking into consideration the correlation between the lutein in the blood and breast milk and the reduction of its levels, similar to all carotenoids, in milk, after 6 days from birth, there is already an important contribution of nutriments high in lutein during breast feeding. Such diet enriched in lutein is particularly important especially for the mothers of premature babies or babies having a small body weight when born. In fact, premature babies and underweight babies need more nutritive essential substances for a fast grow. These babies have not benefit from the contribution of highly nutritive and energetic substances transferred from their mothers during the last weeks of pregnancy. Also, the gastrointestinal and renal functions which are not completely developed reduce the absorption and withhold of important micronutrients, amongst which important antioxidants that protect the newborn from the exposure to high level of free radicals produced excessively at birth and several times as a result of the resuscitation techniques used. Breast feeding is important for the antioxidant contribution to the protection of the newborn and the nutritional state of the mother has subsequently an essential part because it influences the nutrition of the newborn, especially concerning certain solvable nutritive elements, such as lutein and zeaxanthin.

In the literature are already present researches and results with the use of lutein / zeaxanthin in the newborn.

The recent Gong's work has evaluated the role of lutein / zeaxanthin comparing the data obtained from various studies, including those of Romagnoli, Dani and Manzoni. Furthermore, thanks to RCT analysis of Rubin on the subject, investigators concluded that lutein / zeaxanthin is well tolerated and well absorbed from preterm infants also after oral administration.

The extremely interesting result that has emerged although not statistically significant (probably due to the small sample) is that supplementation with lutein / zeaxanthin reduced the incidence and severity of ROP.

This protocol is born from the idea that given the interesting results of earlier work is considered important to deepen a dosage of at least 1 ml / kg equal to 0,5 mg of lutein and 0.05 mg of zeaxanthin.

The evaluation of the key markers for oxidative stress is necessary along with the study of the biological antioxidant potential (BPT) and total hydroperoxide (TH) during and after treatment.

Already in a previous work, S. Perrone and M. Longini have demonstrated a reduction of the free radicals in term infants, during and after administration of lutein / zeaxanthin by determination of the BTP and TH.

Preparations based on lutein and zeaxanthin have never revealed on humans negative or harmful effects after administration, or to the gastrointestinal or systemic level. In recent studies there were not reported adverse phenomena after administrating 20 mg/day of lutein or zeaxanthin for a period of 6 months, or interactions with other liposoluble nutritive elements.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a body weight at birth ≤ 1.500 grams and/or gestational age ≤ 32 weeks
* Male and female newborns
* Newborns whose parents want to sign the informed consent
* Informed consent

Exclusion Criteria:

* Informed consent is not signed
* Infants with a body weight at birth ≥ 1.500 gramms and/or gestational age > 32 weeks
* Infants hospitalized after 36 hours of life
* Infants with Ophthalmologic diseases
* Infants with severe malformations

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-10-11 (Estimated); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Change of the lutein's antioxidant power, after early oral administration in premature newborns | 0 day - 15 days - 30 days
  Biological antioxidant potential (micromol/L) will be analyzed as marker of the antioxidant power. This marker will be tested at birth (0 day) by blood sampling from umbilical vein, while at 15 days and 30 days by peripheral blood
Change of the premature newborns' oxidative stress, after early oral administration of the lutein | 0 day - 15 days - 30 days
  Total hydroperoxide (Ucarr) will be analyzed as marker of the oxidative stress. This marker will be tested at birth (0 day) by blood sampling from umbilical vein, while at 15 days and 30 days by peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Sara Magnanelli, M.D., Study Chair — Sooft Italia; Giuseppe De Bernardo, M.D., Principal Investigator — Sooft Italia
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Padova, Padua, Italia
  - Azienda Ospedaliera Le Scotte Siena, Siena, Italia
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - University Hospital Perugia, Perugia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorenzoni F, Giampietri M, Ferri G, Lunardi S, Madrigali V, Battini L, Boldrini A, Ghirri P. Lutein administration to pregnant women with gestational diabetes mellitus is associated to a decrease of oxidative stress in newborns. Gynecol Endocrinol. 2013 Oct;29(10):901-3. doi: 10.3109/09513590.2013.808329. Epub 2013 Jun 28. PMID 23808391
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Gerardi G, Usberti M, Martini G, Albertini A, Sugherini L, Pompella A, Di LD. Plasma total antioxidant capacity in hemodialyzed patients and its relationships to other biomarkers of oxidative stress and lipid peroxidation. Clin Chem Lab Med. 2002 Feb;40(2):104-10. doi: 10.1515/CCLM.2002.019. PMID 11939481
- [Background] Benzie IF, Strain JJ. The ferric reducing ability of plasma (FRAP) as a measure of "antioxidant power": the FRAP assay. Anal Biochem. 1996 Jul 15;239(1):70-6. doi: 10.1006/abio.1996.0292. PMID 8660627
- [Background] Cohen, J. (1969). Statistical power analysis for the behavioural sciences. New York: Academic Press
- [Result] Shao A, Hathcock JN. Risk assessment for the carotenoids lutein and lycopene. Regul Toxicol Pharmacol. 2006 Aug;45(3):289-98. doi: 10.1016/j.yrtph.2006.05.007. Epub 2006 Jun 30. PMID 16814439
- [Result] Khachik F, London E, de Moura FF, Johnson M, Steidl S, Detolla L, Shipley S, Sanchez R, Chen XQ, Flaws J, Lutty G, McLeod S, Fowler B. Chronic ingestion of (3R,3'R,6'R)-lutein and (3R,3'R)-zeaxanthin in the female rhesus macaque. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5476-86. doi: 10.1167/iovs.06-0194. PMID 17122139
- [Result] Khachik F, de Moura FF, Chew EY, Douglass LW, Ferris FL 3rd, Kim J, Thompson DJ. The effect of lutein and zeaxanthin supplementation on metabolites of these carotenoids in the serum of persons aged 60 or older. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5234-42. doi: 10.1167/iovs.06-0504. PMID 17122108
- [Result] Trevithick-Sutton CC, Foote CS, Collins M, Trevithick JR. The retinal carotenoids zeaxanthin and lutein scavenge superoxide and hydroxyl radicals: a chemiluminescence and ESR study. Mol Vis. 2006 Sep 30;12:1127-35. PMID 17093397
- [Result] Thurmann PA, Schalch W, Aebischer JC, Tenter U, Cohn W. Plasma kinetics of lutein, zeaxanthin, and 3-dehydro-lutein after multiple oral doses of a lutein supplement. Am J Clin Nutr. 2005 Jul;82(1):88-97. doi: 10.1093/ajcn.82.1.88. PMID 16002805
- [Result] Rajendran V, Pu YS, Chen BH. An improved HPLC method for determination of carotenoids in human serum. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Sep 25;824(1-2):99-106. doi: 10.1016/j.jchromb.2005.07.004. PMID 16046287
- [Result] During A, Dawson HD, Harrison EH. Carotenoid transport is decreased and expression of the lipid transporters SR-BI, NPC1L1, and ABCA1 is downregulated in Caco-2 cells treated with ezetimibe. J Nutr. 2005 Oct;135(10):2305-12. doi: 10.1093/jn/135.10.2305. PMID 16177187
- [Result] Reboul E, Abou L, Mikail C, Ghiringhelli O, Andre M, Portugal H, Jourdheuil-Rahmani D, Amiot MJ, Lairon D, Borel P. Lutein transport by Caco-2 TC-7 cells occurs partly by a facilitated process involving the scavenger receptor class B type I (SR-BI). Biochem J. 2005 Apr 15;387(Pt 2):455-61. doi: 10.1042/BJ20040554. PMID 15554873
- [Result] Lutein and zeaxanthin. Monograph. Altern Med Rev. 2005 Jun;10(2):128-35. No abstract available. PMID 15989382
- [Result] Krinsky NI, Landrum JT, Bone RA. Biologic mechanisms of the protective role of lutein and zeaxanthin in the eye. Annu Rev Nutr. 2003;23:171-201. doi: 10.1146/annurev.nutr.23.011702.073307. Epub 2003 Feb 27. PMID 12626691
- [Result] Tyssandier V, Reboul E, Dumas JF, Bouteloup-Demange C, Armand M, Marcand J, Sallas M, Borel P. Processing of vegetable-borne carotenoids in the human stomach and duodenum. Am J Physiol Gastrointest Liver Physiol. 2003 Jun;284(6):G913-23. doi: 10.1152/ajpgi.00410.2002. Epub 2003 Jan 10. PMID 12736146
- [Result] Cardinault N, Gorrand JM, Tyssandier V, Grolier P, Rock E, Borel P. Short-term supplementation with lutein affects biomarkers of lutein status similarly in young and elderly subjects. Exp Gerontol. 2003 May;38(5):573-82. doi: 10.1016/s0531-5565(03)00039-1. PMID 12742535
- [Result] Krinsky NI. Possible biologic mechanisms for a protective role of xanthophylls. J Nutr. 2002 Mar;132(3):540S-542S. doi: 10.1093/jn/132.3.540S. PMID 11880589
- [Result] Granado F, Olmedilla B, Blanco I. Nutritional and clinical relevance of lutein in human health. Br J Nutr. 2003 Sep;90(3):487-502. doi: 10.1079/bjn2003927. PMID 14513828
- [Result] Giuseppe Buonocore, Monica Tei, Serafina Perrone. Lutein as protective agent against neonatal oxidative stress. Journal of Pediatric and Neonatal Individualized Medicine 2014;3(2):e030244.
- [Result] Perrone S, Tei M, Longini M, Santacroce A, Turrisi G, Proietti F, Felici C, Picardi A, Bazzini F, Vasarri P, Buonocore G. Lipid and protein oxidation in newborn infants after lutein administration. Oxid Med Cell Longev. 2014;2014:781454. doi: 10.1155/2014/781454. Epub 2014 Apr 30. PMID 24876916
- [Result] Perrone S, Longini M, Marzocchi B, Picardi A, Bellieni CV, Proietti F, Rodriguez A, Turrisi G, Buonocore G. Effects of lutein on oxidative stress in the term newborn: a pilot study. Neonatology. 2010;97(1):36-40. doi: 10.1159/000227291. Epub 2009 Jul 7. PMID 19590244
- [Result] Shoji H, Koletzko B. Oxidative stress and antioxidant protection in the perinatal period. Curr Opin Clin Nutr Metab Care. 2007 May;10(3):324-8. doi: 10.1097/MCO.0b013e3280a94f6d. PMID 17414502
- [Result] Fokkelman K, Haase E, Stevens J, Idikio H, Korbutt G, Bigam D, Cheung PY. Tissue-specific changes in glutathione content of hypoxic newborn pigs reoxygenated with 21% or 100% oxygen. Eur J Pharmacol. 2007 May 7;562(1-2):132-7. doi: 10.1016/j.ejphar.2007.01.057. Epub 2007 Feb 8. PMID 17349991
- [Result] Franco MC, Akamine EH, Reboucas N, Carvalho MH, Tostes RC, Nigro D, Fortes ZB. Long-term effects of intrauterine malnutrition on vascular function in female offspring: implications of oxidative stress. Life Sci. 2007 Jan 30;80(8):709-15. doi: 10.1016/j.lfs.2006.10.028. Epub 2006 Nov 11. PMID 17157880
- [Result] Mercer JS, Erickson-Owens DA, Graves B, Haley MM. Evidence-based practices for the fetal to newborn transition. J Midwifery Womens Health. 2007 May-Jun;52(3):262-72. doi: 10.1016/j.jmwh.2007.01.005. PMID 17467593
- [Result] Kopsell DA, Lefsrud MG, Kopsell DE, Wenzel AJ, Gerweck C, Curran-Celentano J. Spinach cultigen variation for tissue carotenoid concentrations influences human serum carotenoid levels and macular pigment optical density following a 12-week dietary intervention. J Agric Food Chem. 2006 Oct 18;54(21):7998-8005. doi: 10.1021/jf0614802. PMID 17032001
- [Result] Fanaris, Bel BO, Guidettic E et al. Ruolo della Luteina nella prevenzione delle patologie oculari nel neonato. Rivista Italiana di Medicina Pediatrica 2006;numero speciale:51-53
- [Result] Kvansakul J, Rodriguez-Carmona M, Edgar DF, Barker FM, Kopcke W, Schalch W, Barbur JL. Supplementation with the carotenoids lutein or zeaxanthin improves human visual performance. Ophthalmic Physiol Opt. 2006 Jul;26(4):362-71. doi: 10.1111/j.1475-1313.2006.00387.x. PMID 16792735
- [Result] Rodriguez-Carmona M, Kvansakul J, Harlow JA, Kopcke W, Schalch W, Barbur JL. The effects of supplementation with lutein and/or zeaxanthin on human macular pigment density and colour vision. Ophthalmic Physiol Opt. 2006 Mar;26(2):137-47. doi: 10.1111/j.1475-1313.2006.00386.x. PMID 16460314
- [Result] Provis JM, Penfold PL, Cornish EE, Sandercoe TM, Madigan MC. Anatomy and development of the macula: specialisation and the vulnerability to macular degeneration. Clin Exp Optom. 2005 Sep;88(5):269-81. doi: 10.1111/j.1444-0938.2005.tb06711.x. PMID 16255686
- [Result] Yanoff M and Duker i.S (2005) "Ophthalmology" Edizione italiana ed 2003 ristampa 2005, Antonio Delfino Editore medicina-scienze, volume 1, cap 1.3
- [Result] Santosa S, Jones PJ. Oxidative stress in ocular disease: does lutein play a protective role? CMAJ. 2005 Oct 11;173(8):861-2. doi: 10.1503/cmaj.1031425. No abstract available. PMID 16217103
- [Result] van Leeuwen R, Boekhoorn S, Vingerling JR, Witteman JC, Klaver CC, Hofman A, de Jong PT. Dietary intake of antioxidants and risk of age-related macular degeneration. JAMA. 2005 Dec 28;294(24):3101-7. doi: 10.1001/jama.294.24.3101. PMID 16380590
- [Result] Schweigert FJ, Bathe K, Chen F, Buscher U, Dudenhausen JW. Effect of the stage of lactation in humans on carotenoid levels in milk, blood plasma and plasma lipoprotein fractions. Eur J Nutr. 2004 Feb;43(1):39-44. doi: 10.1007/s00394-004-0439-5. Epub 2004 Jan 6. PMID 14991268
- [Result] Jewell VC, Mayes CB, Tubman TR, Northrop-Clewes CA, Thurnham DI. A comparison of lutein and zeaxanthin concentrations in formula and human milk samples from Northern Ireland mothers. Eur J Clin Nutr. 2004 Jan;58(1):90-7. doi: 10.1038/sj.ejcn.1601753. PMID 14679372
- [Result] Nolan J, O'Donovan O, Kavanagh H, Stack J, Harrison M, Muldoon A, Mellerio J, Beatty S. Macular pigment and percentage of body fat. Invest Ophthalmol Vis Sci. 2004 Nov;45(11):3940-50. doi: 10.1167/iovs.04-0273. PMID 15505040
- [Result] Richer S, Stiles W, Statkute L, Pulido J, Frankowski J, Rudy D, Pei K, Tsipursky M, Nyland J. Double-masked, placebo-controlled, randomized trial of lutein and antioxidant supplementation in the intervention of atrophic age-related macular degeneration: the Veterans LAST study (Lutein Antioxidant Supplementation Trial). Optometry. 2004 Apr;75(4):216-30. doi: 10.1016/s1529-1839(04)70049-4. PMID 15117055
- [Result] Vento M, Asensi M, Sastre J, Lloret A, Garcia-Sala F, Vina J. Oxidative stress in asphyxiated term infants resuscitated with 100% oxygen. J Pediatr. 2003 Mar;142(3):240-6. doi: 10.1067/mpd.2003.91. PMID 12640369
- [Result] Broekmans WM, Berendschot TT, Klopping-Ketelaars IA, de Vries AJ, Goldbohm RA, Tijburg LB, Kardinaal AF, van Poppel G. Macular pigment density in relation to serum and adipose tissue concentrations of lutein and serum concentrations of zeaxanthin. Am J Clin Nutr. 2002 Sep;76(3):595-603. doi: 10.1093/ajcn/76.3.595. PMID 12198005
- [Result] Gossage CP, Deyhim M, Yamini S, Douglass LW, Moser-Veillon PB. Carotenoid composition of human milk during the first month postpartum and the response to beta-carotene supplementation. Am J Clin Nutr. 2002 Jul;76(1):193-7. doi: 10.1093/ajcn/76.1.193. PMID 12081834
- [Result] Jewell VC, Northrop-Clewes CA, Tubman R, Thurnham DI. Nutritional factors and visual function in premature infants. Proc Nutr Soc. 2001 May;60(2):171-8. doi: 10.1079/pns200089. PMID 11681632
- [Result] Vento M, Asensi M, Sastre J, Garcia-Sala F, Pallardo FV, Vina J. Resuscitation with room air instead of 100% oxygen prevents oxidative stress in moderately asphyxiated term neonates. Pediatrics. 2001 Apr;107(4):642-7. doi: 10.1542/peds.107.4.642. PMID 11335737
- [Result] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Result] Sommerburg O, Meissner K, Nelle M, Lenhartz H, Leichsenring M. Carotenoid supply in breast-fed and formula-fed neonates. Eur J Pediatr. 2000 Jan-Feb;159(1-2):86-90. doi: 10.1007/pl00013811. PMID 10653337
- [Result] Kiely M, Cogan PF, Kearney PJ, Morrissey PA. Concentrations of tocopherols and carotenoids in maternal and cord blood plasma. Eur J Clin Nutr. 1999 Sep;53(9):711-5. doi: 10.1038/sj.ejcn.1600838. PMID 10509767
- [Result] Yeum KJ, Ferland G, Patry J, Russell RM. Relationship of plasma carotenoids, retinol and tocopherols in mothers and newborn infants. J Am Coll Nutr. 1998 Oct;17(5):442-7. doi: 10.1080/07315724.1998.10718791. PMID 9791840
- [Result] Oostenbrug GS, Mensink RP, Al MD, van Houwelingen AC, Hornstra G. Maternal and neonatal plasma antioxidant levels in normal pregnancy, and the relationship with fatty acid unsaturation. Br J Nutr. 1998 Jul;80(1):67-73. doi: 10.1017/s0007114598001780. PMID 9797645
- [Result] Bonn D. Keeping the stork at bay until the time is right. Lancet. 1998 Feb 21;351(9102):576. doi: 10.1016/S0140-6736(05)78569-X. No abstract available. PMID 9492791
- [Result] Sommerburg O, Keunen JE, Bird AC, van Kuijk FJ. Fruits and vegetables that are sources for lutein and zeaxanthin: the macular pigment in human eyes. Br J Ophthalmol. 1998 Aug;82(8):907-10. doi: 10.1136/bjo.82.8.907. PMID 9828775
- [Result] Jackson JG, Eric L, Lien A, Sharon J, White B, Nicholas J, Bruns C, Charles F, Kuhlman A. Major carotenoids in mature human milk: longitudinal and diurnal patterns. The Journal of Nutritional Biochemistry 1998 Jan;9(1):2-7.
- [Result] Khachik F, Spangler CJ, Smith JC Jr, Canfield LM, Steck A, Pfander H. Identification, quantification, and relative concentrations of carotenoids and their metabolites in human milk and serum. Anal Chem. 1997 May 15;69(10):1873-81. doi: 10.1021/ac961085i. PMID 9164160
- [Result] Landrum JT, Bone RA, Joa H, Kilburn MD, Moore LL, Sprague KE. A one year study of the macular pigment: the effect of 140 days of a lutein supplement. Exp Eye Res. 1997 Jul;65(1):57-62. doi: 10.1006/exer.1997.0309. PMID 9237865
- [Result] Leung AK, Siu TO, Chiu AS, Robson WL, Larsen TE. Serum carotene concentrations in normal infants and children. Clin Pediatr (Phila). 1990 Oct;29(10):575-8; discussion 579-80. doi: 10.1177/000992289002901004. PMID 2253431
- [Result] Nakamura H, Lee Y, Uetani Y, Kitsunezuka Y, Shimabuku R, Matsuo T. Effects of phototherapy on serum unbound bilirubin i icteric newborn infants. Biol Neonate. 1981;39(5-6):295-9. doi: 10.1159/000241451. PMID 7260214
- [Result] Alberti A, Bolognini L, Macciantelli D, et al. The radical cation of N,N-dimethyl-para-phenylendiamine: a possible indicator of oxidative stress in biological samples. Res Chem Intermed 2000; 26:253-267

DOCUMENTS (2):
  • Informed Consent Form (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03340103/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03340103/Prot_SAP_001.pdf